CLINICAL TRIAL: NCT05775887
Title: A PHASE 1 RANDOMIZED, ACTIVE-CONTROLLED, DOUBLEBLIND, SINGLE CENTRE STUDY TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF AN ADJUVANTED SARS-CoV-2 UQSC2 PROTEIN SUBUNIT VACCINE IN HEALTHY ADULTS, AGED 18 TO 50 YEARS.
Brief Title: A FIRST IN HUMAN TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF SARS-CoV-2 UQSC2 VACCINE IN HEALTHY ADULTS.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Queensland (Other)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UQ-2-UQSC2
Record Dates: First submitted 2023-03-08; First posted 2023-03-20 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: SARS-CoV-2 infection; vaccine
MeSH Terms: conditions — COVID-19 | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UQSC2 vaccine (Experimental): 15mcg of UQSC2 (SARS-CoV-2 Sclamp2 antigen) adjuvanted with MF59
  Interventions: Biological: UQSC2 Vaccine
- NVX-CoV2373 vaccine (Active Comparator): 5 mcg SARS-CoV-2 spike protein adjuvanted with Matrix-M
  Interventions: Biological: NVX-CoV2373 vaccine

INTERVENTIONS:
Biological: UQSC2 Vaccine — Subjects will be assigned to treatment group (UQSC2 or NVX-CoV2373) via randomisation. Each treatment group will receive a single dose of either UQSC2 or NVX-CoV2373. The Study will be unblinded after Day 29, to enable subjects who received the investigational vaccine (UQSC2 vaccine) to seek vaccination with a TGA (Therapeutic Goods Administration) approved COVID-19 booster vaccine if indicated by public health authorities.
  Arms: UQSC2 vaccine
Biological: NVX-CoV2373 vaccine — Subjects will be assigned to treatment group (UQSC2 or NVX-CoV2373) via randomisation. Each treatment group will receive a single dose of either UQSC2 or NVX-CoV2373
  Arms: NVX-CoV2373 vaccine

SUMMARY:
This will be a single centre, Phase 1, First-In-Human , Randomized, Active-controlled (2- arm) Double-blind, single dose, parallel design study. The study will be conducted in a young healthy adult population aged ≥ 18 - ≤ 50 years. This study will consist of a single cohort of 70 subjects (35 receiving a single dose of UQSC2 vaccine and 35 subjects receiving a single dose of a TGA (Therapeutic Goods Administration) registered SARS-CoV-2 vaccine NVX-CoV2373).

DETAILED DESCRIPTION:
Approximately 70 healthy adult males or non-pregnant females, ≥18 years - ≤ 50 years of age, non-smokers and social smokers (defined as the equivalent or fewer than 10 cigarettes per week), with BMI >18.0 and <34.0 kg/m2, will be recruited for participation in this study.

All participants must have completed a primary SARS-CoV-2 vaccination series with one of two authorised mRNA SARS-CoV-2 vaccines (Pfizer/BioNTech or Moderna) and have received at least one booster dose of the Pfizer or Moderna SARS-CoV-2 vaccine at least 3 months prior to study entry, and will have not had a history of COVID-19 or virologically confirmed SARS-CoV-2 infection in the past 3 months, or will not have ongoing sequelae from a past COVID-19 infection.

Subjects will be assigned to treatment group (UQSC2 or NVX-CoV2373) via randomisation.

Each treatment group will receive a single dose of either UQSC2 or NVXCoV2373.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or non-pregnant female, ≥18 and ≤50 years of age, with BMI ≥18 and ≤ 34.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
2. Healthy as defined by:

   1. The absence of clinically significant illness and surgery within 28 days prior to dosing. Subjects displaying signs or symptoms of an acute and/or febrile illness within 24 hours pre-dose (at least 3 symptom-free pre-dose days required) will be carefully evaluated for upcoming illness/disease. Inclusion of pre-dosing is at the discretion of the Investigator, and the subject may have their scheduled dosing postponed until the condition resolves.
   2. The absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, haematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
3. Non-smokers or social smokers (defined as the equivalent or fewer than 10 cigarettes per week). Ex-heavy smokers (heavy smoking is defined as the equivalent of 25 or more cigarettes per day) may be admitted if they have quit or reduced their cigarette intake to the defined level of social smoking, for a period of at least 12 months. Ex-moderate level smokers (i.e. >10 per week but <25 per day) may be admitted if they have quit or reduced their cigarette intake to the defined level of social smoking, for a period of at least 6 months.
4. All women of child bearing potential (WOCBP) and men must refrain from sperm/egg donation and must be able and willing to use at least 1 highly effective method of contraception commencing at least 28 days prior to vaccine administration and for 3 months after vaccine administration. Subjects in same sex relationships must be able and willing to refrain from sperm/egg donation for 3 months after vaccine administration. A female subject is considered to be a WOCBP following menarche and until she is in a post-menopausal state for 12 consecutive months (without an alternative medical cause) or otherwise permanently sterile (for which acceptable methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy). A follicle-stimulating hormone (FSH) test may be used to confirm a post-menopausal state. Examples of acceptable methods of contraceptive methods (for female subjects and female partners of male subjects) to be used throughout the study include

   1. Use of hormonal contraceptives, started at at least 28 days prior to study treatment administration and must agree to use the same hormonal contraceptive throughout the study;
   2. Use of an intra-uterine contraceptive device, placed at at least 28 days prior to study treatment administration;
   3. Use of a diaphragm, started at least 28 days prior to study treatment administration;
   4. Use of condoms for male subjects whose partners are pregnant to ensure that the foetus is not exposed to the study vaccine;
   5. Sterile male partner (vasectomized since at least 6 months prior to study treatment administration)
   6. True abstinence, defined as no sexual intercourse with a male partner, (for heterosexual couples) from the time of enrollment and at for at least 28 days prior to study treatment administration and for at least the duration of the study. Periodic abstinence and withdrawal are not acceptable methods.
5. Must meet the following COVID-19 vaccination status:

   1. Have completed a primary SARS-CoV-2 vaccination series with either the Pfizer or Moderna COVID-19 vaccine, and
   2. Have received at least one booster dose of the Pfizer or Moderna SARS-CoV-2 vaccine at least 3 months prior to study entry.
6. WOCBP must return a negative urine pregnancy test prior to receiving the study treatment.
7. Male subjects (including men who have had a vasectomy) with a pregnant partner, a female partner not of childbearing potential, or a same sex partner, must agree to use a condom from study treatment administration until at least 90 days after the last study treatment administration.
8. Must be willing to refrain from blood (and plasma) donation throughout study participation.
9. Must be able to attend all visits for the duration of the study and comply with all study procedures according to the study schedule.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

1. Any clinically significant abnormality or vital sign abnormality at physical examination (including baseline resting average high blood pressure [average systolic blood pressure ≥140 mmHg or resting average diastolic blood pressure ≥90 mmHg or high random blood sugar [nonfasting]), clinically significant abnormal laboratory test results or positive test for HIV, hepatitis B, or hepatitis C found during medical screening.
2. Any acute or chronic ongoing illness which, in the judgement of the investigator, may preclude the subject's participation. Subjects who have a chronic condition that is stable and controlled and otherwise healthy should not be excluded. Within at least the past 3 months must NOT have received another COVID-19 vaccine.
3. Persons who received another COVID-19 vaccine within the past 3 months prior to dosing.
4. Persons who received a primary vaccination series and or a booster vaccination dose of a non-mRNA COVID-19 vaccine (ie Matrix M adjuvanted COVID-19 vaccine, Novavax).
5. Persons who have a history of COVID-19 or virologically confirmed SARS-CoV-2 infection in the past 3 months.
6. Persons with a history of COVID-19 with ongoing sequelae.
7. Persons with a history of myocarditis and/or pericarditis.
8. Positive pregnancy, urine drug screen, or alcohol breath test at screening.
9. Known history of allergic reactions or hypersensitivity to any vaccine, or to any excipient in the formulation (including the adjuvants: MF59C.1 and Matrix-M).
10. Presence of a known, or suspected, impairment of the immune system including, but not limited to, HIV, autoimmune disorders, immunosuppressant therapy, and diabetes mellitus.
11. History of a known, or suspected, respiratory system disorder including, but not limited to, cystic fibrosis, reactive airway disease, emphysema, chronic bronchitis, chronic obstructive pulmonary disease (COPD), or asthma, excluding childhood asthma.
12. History of significant alcohol abuse within 12 months prior to screening.
13. Positive test for drugs of abuse (such as marijuana/ tetrahydrocannabinol [THC] products, amphetamine, methamphetamine, methadone, barbiturates, benzodiazepines, cocaine, opiates, methylenedioxymethamphetamine [MDMA], or phencyclidine [PCP]) at screening, prior to dosing, or a history of drug abuse within 12months prior to screening.
14. Participation in a clinical research study involving the administration of an investigational, or marketed, drug or device within 30 days prior to receiving the treatment administration, or administration of a biological product in the context of a clinical research study within 90 days prior to dosing, or concomitant participation in an investigational study involving drug, vaccine, or device administration, or intent to participate in another clinical study at any time during the conduct of the study.
15. Use of medications for the timeframes specified below, (except for hormonal contraceptives and medications exempted by the Investigator on a case-by-case basis) because they are judged to interfere with subject safety e.g., topical drug products without significant systemic absorption are permissible:

    1. A new, or a change in a prescription medication within 14 days prior to treatment administration;
    2. Any medication, or treatments, that may affect the immune system such as allergy injections, immunoglobulin, interferon, immunomodulators, cytotoxic drugs, or other drugs are known to be frequently associated with significant major organ toxicity within 90 days prior to enrolment;
    3. Any registered vaccine administered within 30 days prior to enrolment in the study, or who plan to receive any non-study vaccines within 28 days of the study vaccine
    4. Any other investigational coronavirus vaccine i.e. SARS-CoV-1, SARS-CoV-2, MERS etc. at any time prior to, or during, the study.
    5. Over-the-counter products within 7 days prior to dosing, with the exception of the occasional use of paracetamol (up to 2 g daily) and standard dose vitamins.
16. Donation of plasma within 7 days prior to dosing. Donation or loss of blood (excluding volume drawn at screening) of 50 mL to 499 mL of blood within 30 days, or more than 499 mL within 56 days prior to dosing.
17. Receipt of blood products within 2 months prior to vaccine administration (Day 1), or planned receipt of blood products during the study period (Screening through Day 29).
18. Breast-feeding subjects, or subjects who plan to breastfeed from the time of the vaccination through 60 days after the treatment administration.
19. Presence of tattoos, scarring, skin discolouration, or any other skin disturbances at the injection site which, in the opinion of the Investigator, may inhibit the ability to effectively perform an injection site assessment.
20. Employee or immediate relative of an employee of the clinical site, any of its affiliates or partners, or Syneos Health.
21. Employees of the specific team at the University of Queensland responsible for manufacturing and managing the IP (Investigational Product) or their immediate relatives.
22. Any reason that, in the opinion of the Investigator, would interfere with the primary study objectives or prevent the subject from participating in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Frequency, duration, and intensity of solicited local adverse events (AEs) | [Time Frame: Day 1-7]
  Frequency, duration, and intensity of solicited local adverse events (AEs), including pain, redness, and induration for 7 days following vaccination.
Frequency, duration, and intensity of solicited systemic adverse events (AEs) | [Time Frame: Day 1-7]
  Frequency, duration, and intensity of solicited systemic adverse events (AEs), including fever, nausea, chills,diarrhoea, headache, fatigue, and myalgia for 7 days following vaccination.
Frequency, duration, and intensity of solicited systemic adverse events (AEs) | [Time Frame: Day 1-29]
  Frequency, duration, and intensity of solicited systemic adverse events (AEs)
Frequency of Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest and any AEs leading to study withdrawal at any time | [Time Frame: Dat 1-183]
  Frequency of Serious Adverse Events (SAEs), Medically Attended Adverse Events (MAAEs), Adverse Events of Special Interest (AESIs, namely myocarditis, pericarditis, anaphylaxis, thrombocytopaenia, Acute disseminated encephalomyelitis (ADEM) and Guillain-Barre Syndrome (GBS) and any AEs leading to study withdrawal at any time during the study through to Day 183.
Geometric Mean Titres (GMT) of the serum NAb (Neutralising Antibody) titres to matched SARS-CoV-2 (prototypic strain) by microneutralisation (MN) assay. | [Time Frame: At Day 29]
  Geometric Mean Titres (GMT) of the serum NAb titres to matched SARS-CoV-2 (prototypic strain) by microneutralisation (MN) assay at Day 29 (28 days after vaccination) relative to day 1 (pre-dosing), compared to NVXCoV2373.
Seroresponse rate (SRR), where seroresponse is defined as ≥ 4-fold rise from pre-vaccination, Day 1) by MN assay to matched SARS-CoV-2 (prototypic strain). | [Time Frame: At Day 29]
  Seroresponse rate (SRR), where seroresponse is defined as ≥ 4-fold rise from pre-vaccination, Day 1) by MN assay to matched SARS-CoV-2 (prototypic strain) at Day 29 compared to NVX-CoV2373.

SECONDARY OUTCOMES:
GMT of the serum antibody response by SARS-CoV-2 Spike antigen specific ELISA | [Time Frame: At Day 29]
  GMT of the serum antibody response by SARS-CoV-2 Spike antigen specific ELISA at Day 29 (28 days after booster dose) relative to Day 1 (pre-booster dosing), compared to NVX-CoV2373.
Seroresponse rate (SRR, where seroresponse is defined as ≥ 4-fold rise from pre-vaccination, Day 1) by ELISA | [Time Frame: At Days 15, 29, 91 and 183]
  Seroresponse rate (SRR, where seroresponse is defined as ≥ 4-fold rise from pre-vaccination, Day 1) by ELISA at Days 15, 29, 91 and 183, compared to NVX-CoV2373.
SRR by MN assay at Days 15, 29, 91 and183, compared to NVX-CoV2373 | [Time Frame: At Days 15, 29, 91 and 183]
  SRR by MN assay at Days 15, 29, 91 and183, compared to NVX-CoV2373.
GMT to the SARS-CoV-2 Spike by antigen specific ELISA | [Time Frame: At Days 1,15, 29, 91 and 183]
  GMT to the SARS-CoV-2 Spike by antigen specific ELISA at Days 1, 15, 29, 91 and183, compared to NVX-CoV2373.
GMT of the serum NAb titres to matched SARS-CoV-2 (prototypic strain) by MN assay | [Time Frame: At Days 1,15, 29, 91 and 183]
  GMT of the serum NAb titres to matched SARS-CoV-2 (prototypic strain) by MN assay at Days 1, 15, 29, 91 and183, compared to NVX-CoV2373.

CONTACTS AND LOCATIONS:
Overall Officials: Kristi Mclendon, Principal Investigator — Nucleus Network Pty Ltd Brisbane
Locations (1):
- QPharm Pty.Ltd. (Nucleus Network Brisbane), Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No
Study results will be published

REFERENCES:
- [Derived] Chappell KJ, Mordant FL, Amarilla AA, Modhiran N, Liang B, Li Z, Lackenby JA, Jaberolansar N, O'Donnell J, Kienzle V, Kommajosyula V, Tardiota N, Bennet JK, Henderson CL, Dalrymple RL, Goh J, Hoger K, Gillard M, Jones ML, Hughes K, Hughes B, Barnes J, Reading PC, Ranasinghe C, Subbarao K, Munro TP, Young PR, Watterson D. Safety and immunogenicity of a SARS-CoV-2 spike, subunit vaccine stabilised in the prefusion conformation by second generation Molecular Clamp evaluated in adults aged 18-55 years: a randomised, double-blind, active comparator, Phase I trial. J Infect Dis. 2025 Nov 25:jiaf568. doi: 10.1093/infdis/jiaf568. Online ahead of print. PMID 41285172